CLINICAL TRIAL: NCT05607316
Title: Metformin as a Novel Treatment for Vitiligo by Targeting CD8+ T Cell Metabolism
Brief Title: Evaluating the Efficacy and Safety of Metformin in Vitiligo
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to secure funding.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, John Harris, Chair, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000630
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Vitiligo
Keywords: vitiligo; metformin; systemic treatment; stable vitiligo; segmental vitiligo; non-segmental vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Open-label (unmasked) study
Masking Description: Open-label (unmasked)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Metformin (Experimental): Treatment with metformin will be started at 500 mg twice daily and increased to 1000 mg twice daily only after they have tolerated the treatment.
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Consistent with previous studies and clinical recommendations, subjects will initiate treatment at metformin 500 mg twice daily and increase to 1000 mg twice daily only after they have tolerated the treatment (details below).
  Study Visit 1 (Week 1) - Study Visit 2 (Week 2) Subjects will be directed to take metformin 500 mg twice daily.
  Study Visit 2 (Week 2) - Study Visit 5 (Week 24) If initial metformin dose is tolerated, subjects will be directed to increase the dose to 1000 mg by mouth twice daily for the remainder of the study.
  Other Names: Glucophage; Glumetza; Riomet

SUMMARY:
Metformin modulates metabolism in multiple cell types and is currently used to reduce glucose levels and insulin resistance in diabetic patients. The investigators hypothesize that oral metformin can regulate the metabolism of CD8+ T cells, reduce their cytotoxic activity and thus serve as a novel treatment for vitiligo.

DETAILED DESCRIPTION:
Metformin modulates metabolism in multiple cell types and is currently used to reduce glucose levels and insulin resistance in diabetic patients. It has been reported that the use of metformin correlated with a lower risk of developing vitiligo, suggesting that metformin could potentially mitigate the disease. The investigators found that treating mouse T cells with metformin during activation reduced their mitochondrial respiration and proliferation, while mice treated with metformin reversed their vitiligo. Therefore, the investigators hypothesize that regulation of CD8+ T cell metabolism in vitiligo patients by metformin will reduce their proliferation and cytotoxic activity, resulting in skin repigmentation and thus serve as a novel treatment.

The investigators plan to treat approximately 30 subjects with stable vitiligo.

Metformin is FDA-approved for use with dosing from 500-2000 mg/day. It has a rare risk of lactic acidosis, which can be meaningful in patients with risk factors such as renal insufficiency. This risk is directly proportional to the dose given; therefore, participants will be started at a lower dose (500 mg twice daily) with follow-up to monitor any arising symptoms. Per current clinical recommendations, participants will only be increased to higher-dose metformin (1000 mg twice daily) if the initial dose is tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years - 100 years of age with stable vitiligo

  * Stable vitiligo is defined as no new spots of depigmentation or expansion of any existing spots for one year;
  * Total body surface area BSA >/= 1%
  * Facial body surface area BSA >/= 0.25%
* Willingness to participate in the study;
* Willingness to undergo suction blistering;
* Non-English speaking adults may be enrolled with the assistance of an interpreter and the use of an IRB-approved short form in the subject's language;
* Informed consent document signed by the subject;

Exclusion Criteria:

* Adults unable to consent (adults lacking capacity);
* Active vitiligo defined by presence of confetti lesions, trichrome lesions, and Koebner's phenomenon;
* Individuals who are not yet adults (infants, children, teenagers);
* Pregnant women and/or breastfeeding, or those who have recently delivered a baby within the past 6 months;
* Prisoners;
* Systemic immunosuppressive medication (oral corticosteroids) within prior 4 weeks;
* Topical steroids within the prior 2 weeks;
* Currently undergoing UVB light therapy or history of light therapy within the past 8 weeks;
* Unable to return for follow-up visits;
* Enrolled in a clinical study of any other investigational drug or device;
* Diabetes, liver disease, or kidney disease;
* Hypoglycemia as defined by fasting blood glucose <70 mg/dL assessed at a fasting study visit;
* Prescription medication or cosmetics containing: retinoids, glycolic acid, salicylic acid, or any other remedies that might affect the healing process. Non-medicated moisturizers are allowed. If the person is unsure, they can bring in any products for our review;
* Self-reported history of chronic alcohol or drug abuse within 12 months prior to screening, or any condition associated with poor compliance as judged by the investigator;
* Any other condition or laboratory value that would, in the professional opinion of the investigators, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Define the different populations of cells by flow cytometry | Week 24
  Determine any change in the subpopulations of CD8+ T cells using CD69 and CD103 for Trm and CD122 (IL15Rb chain) as a marker for long-lived Trm; CD44, CD62L, and CD127 for central and effector memory T cells; and CXCR3 to indicate trafficking of CD8+ T cells.

SECONDARY OUTCOMES:
Define the inflammatory conditions in the lesions | Week 24
  Protein biomarker discovery using Olink® proteomics technology platform (inflammation panel)
Measure the abundance of metabolites with untargeted metabolomics in the blister fluid and cells from non-lesional and lesional areas, and in plasma | Week 24
  Liquid chromatography-mass spectrometry
Vitiligo Area Scoring Index 50% improvement (VASI50) after 6 months of treatment | Week 24
  Assess VASI at baseline and after 3 months of starting treatment.
Face-Vitiligo Area Scoring Index 50% improvement (F-VASI50) after 6 months of treatment | Week 24
  Assess facial VASI at baseline and after 6 months of starting treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John E Harris, MD, PhD, Principal Investigator — Chair, Department of Dermatology
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rashighi M, Agarwal P, Richmond JM, Harris TH, Dresser K, Su MW, Zhou Y, Deng A, Hunter CA, Luster AD, Harris JE. CXCL10 is critical for the progression and maintenance of depigmentation in a mouse model of vitiligo. Sci Transl Med. 2014 Feb 12;6(223):223ra23. doi: 10.1126/scitranslmed.3007811. PMID 24523323
- [Background] Zhang Y, Cai Y, Shi M, Jiang S, Cui S, Wu Y, Gao XH, Chen HD. The Prevalence of Vitiligo: A Meta-Analysis. PLoS One. 2016 Sep 27;11(9):e0163806. doi: 10.1371/journal.pone.0163806. eCollection 2016. PMID 27673680
- [Background] Salzes C, Abadie S, Seneschal J, Whitton M, Meurant JM, Jouary T, Ballanger F, Boralevi F, Taieb A, Taieb C, Ezzedine K. The Vitiligo Impact Patient Scale (VIPs): Development and Validation of a Vitiligo Burden Assessment Tool. J Invest Dermatol. 2016 Jan;136(1):52-8. doi: 10.1038/JID.2015.398. PMID 26763423
- [Background] Linthorst Homan MW, Spuls PI, de Korte J, Bos JD, Sprangers MA, van der Veen JP. The burden of vitiligo: patient characteristics associated with quality of life. J Am Acad Dermatol. 2009 Sep;61(3):411-20. doi: 10.1016/j.jaad.2009.03.022. Epub 2009 Jul 3. PMID 19577331
- [Background] Elbuluk N, Ezzedine K. Quality of Life, Burden of Disease, Co-morbidities, and Systemic Effects in Vitiligo Patients. Dermatol Clin. 2017 Apr;35(2):117-128. doi: 10.1016/j.det.2016.11.002. PMID 28317521
- [Background] Ogg GS, Rod Dunbar P, Romero P, Chen JL, Cerundolo V. High frequency of skin-homing melanocyte-specific cytotoxic T lymphocytes in autoimmune vitiligo. J Exp Med. 1998 Sep 21;188(6):1203-8. doi: 10.1084/jem.188.6.1203. PMID 9743539
- [Background] Frisoli ML, Essien K, Harris JE. Vitiligo: Mechanisms of Pathogenesis and Treatment. Annu Rev Immunol. 2020 Apr 26;38:621-648. doi: 10.1146/annurev-immunol-100919-023531. Epub 2020 Feb 4. PMID 32017656
- [Background] Richmond JM, Bangari DS, Essien KI, Currimbhoy SD, Groom JR, Pandya AG, Youd ME, Luster AD, Harris JE. Keratinocyte-Derived Chemokines Orchestrate T-Cell Positioning in the Epidermis during Vitiligo and May Serve as Biomarkers of Disease. J Invest Dermatol. 2017 Feb;137(2):350-358. doi: 10.1016/j.jid.2016.09.016. Epub 2016 Sep 26. PMID 27686391
- [Background] Sanchez-Rangel E, Inzucchi SE. Metformin: clinical use in type 2 diabetes. Diabetologia. 2017 Sep;60(9):1586-1593. doi: 10.1007/s00125-017-4336-x. Epub 2017 Aug 2. PMID 28770321
- [Background] Agius L, Ford BE, Chachra SS. The Metformin Mechanism on Gluconeogenesis and AMPK Activation: The Metabolite Perspective. Int J Mol Sci. 2020 May 3;21(9):3240. doi: 10.3390/ijms21093240. PMID 32375255
- [Background] Cui Y, Chang L, Wang C, Han X, Mu L, Hao Y, Liu C, Zhao J, Zhang T, Zhang H, Zhang Y, Liu Y, Zhao W, Wang J, Liu X, Sun B, Wang G, Kong Q, Han J, Li H. Metformin attenuates autoimmune disease of the neuromotor system in animal models of myasthenia gravis. Int Immunopharmacol. 2019 Oct;75:105822. doi: 10.1016/j.intimp.2019.105822. Epub 2019 Aug 19. PMID 31437793
- [Background] Tomczynska M, Bijak M, Saluk J. Metformin - The Drug for the Treatment of Autoimmune Diseases; A New Use of a Known Anti-Diabetic Drug. Curr Top Med Chem. 2016;16(19):2223-30. doi: 10.2174/1568026616666160216152324. PMID 26881720
- [Background] Salvatore T, Pafundi PC, Galiero R, Gjeloshi K, Masini F, Acierno C, Di Martino A, Albanese G, Alfano M, Rinaldi L, Sasso FC. Metformin: A Potential Therapeutic Tool for Rheumatologists. Pharmaceuticals (Basel). 2020 Sep 4;13(9):234. doi: 10.3390/ph13090234. PMID 32899806
- [Background] Doyle-Delgado K, Chamberlain JJ, Shubrook JH, Skolnik N, Trujillo J. Pharmacologic Approaches to Glycemic Treatment of Type 2 Diabetes: Synopsis of the 2020 American Diabetes Association's Standards of Medical Care in Diabetes Clinical Guideline. Ann Intern Med. 2020 Nov 17;173(10):813-821. doi: 10.7326/M20-2470. Epub 2020 Sep 1. PMID 32866414
- [Background] Cornell S. Comparison of the diabetes guidelines from the ADA/EASD and the AACE/ACE. J Am Pharm Assoc (2003). 2017 Mar-Apr;57(2):261-265. doi: 10.1016/j.japh.2016.11.005. Epub 2017 Jan 5. PMID 28065547
- [Background] DeFronzo R, Fleming GA, Chen K, Bicsak TA. Metformin-associated lactic acidosis: Current perspectives on causes and risk. Metabolism. 2016 Feb;65(2):20-9. doi: 10.1016/j.metabol.2015.10.014. Epub 2015 Oct 9. PMID 26773926